CLINICAL TRIAL: NCT02164006
Title: A Multi-center Phase I/Ib Study Evaluating the Efficacy and Safety of Brentuximab Vedotin in Combination With TGR-1202, a Novel PI3K Delta Inhibitor, in Patients With Hodgkins Lymphoma
Brief Title: Novel PI3K Delta Inhibitor TGR-1202, in Combination With Brentuximab Vedotin for Hodgkin's Lymphoma Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: TG Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TGR-BV-107
Record Dates: First submitted 2014-06-12; First posted 2014-06-16 (Estimated); Last update posted 2019-10-02 (Actual); Status verified 2019-10

CONDITIONS: Hodgkin's Lymphoma
Keywords: Hodgkin's
MeSH Terms: conditions — Hodgkin Disease | interventions — umbralisib; Brentuximab Vedotin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- TGR-1202 + brentuximab vedotin (Experimental): TGR-1202 oral daily dose in combination with a fixed IV infusion of brentuximab vedotin
  Interventions: Drug: TGR-1202 + brentuximab vedotin

INTERVENTIONS:
Drug: TGR-1202 + brentuximab vedotin — TGR-1202 an oral daily dose with an IV infusion of brentuximab vedotin
  Other Names: brentuximab vedotin: Adcetris

SUMMARY:
The purpose of this study is to evaluate the safety and effectiveness of TGR-1202 in combination with brentuximab vedotin in patients with hodgkin's lymphoma.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of Hodgkin's Lymphoma
* Relapsed or refractory after an autologous stem cell transplant (ASCT) or at least two prior multi-agent chemotherapy regimens in patients not candidates for ASCT
* Eastern Cooperative Oncology Group (ECOG) score of 0 to 2

Exclusion Criteria:

* Any major surgery, chemotherapy or immunotherapy within the last 21 days
* Known hepatitis B virus, hepatitis C virus or HIV infection
* Autologous hematologic stem cell transplant within 3 months of study entry. Patients who had prior Allogeneic hematologic stem cell transplant are excluded

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2014-06-11 (Actual); Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose acceptable for participants | 21 days (1 cycle of therapy)
  To determine the incidence of adverse events, any potential abnormal laboratory results and any dose-limiting toxicities

SECONDARY OUTCOMES:
Overall Response Rate | Up to 1 year
  To assess the overall response rate (ORR) of TGR-1202 in combination with brentuximab vedotin in patients with Hodgkin's lymphoma

OTHER OUTCOMES:
Duration of Response | Up to 1 year
  To evaluate the duration of response of TGR-1202 in combination with brentuximab vedotin

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - TG Therapeutics Investigational Trial Site, Duarte, California
  - TG Therapeutics Investigational Trial Site, San Diego, California
  - TG Therapeutics Investigational Trial Site, Sarasota, Florida
  - TG Therapeutics Investigational Trial Site, Detroit, Michigan